CLINICAL TRIAL: NCT04733053
Title: The POWER Study: Effects of a Physiotherapist-delivered Dietary Weight Loss Program in Addition to Exercise in People with Knee Osteoarthritis Who Have Overweight or Obesity - a Randomised Controlled Trial
Brief Title: Effects of a Physiotherapist-delivered Dietary Weight Loss Program in People with Knee OA Who Have Overweight/obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1261-5151
Record Dates: First submitted 2021-01-13; First posted 2021-02-01 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis; Overweight and Obesity
MeSH Terms: conditions — Osteoarthritis, Knee; Overweight; Obesity | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The components of each treatment arm will be disclosed to participants as we wish to test the interventions under real world conditions whereby consumers are fully informed about the nature of the components before choosing whether or not they wish to participate. The research staff collecting non-self-reported outcome measures (including the primary outcome) will be blinded to group allocation. The staff member collecting laboratory measures at 6 months will be different to the staff member who collects the baseline data. It is not possible to blind physiotherapists as they are providing interventions to both trial arms (in order to ensure physiotherapist-related factors such as personality, clinical practice experience etc are similar across groups and cannot confound results). The person performing the statistical analyses will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diet plus exercise (Experimental): The initial physiotherapy consultation for participants in this group will last 75 minutes, with 30 minutes for the exercise component and 45 minutes for the diet component. Thereafter, consultations will last 50 minutes, with 20 minutes for the exercise component and 30 minutes for the diet component. The exercise component will be the same as that described for the exercise alone group.
  Interventions: Other: Diet plus exercise; Other: Exercise
- Exercise (Active Comparator): Physiotherapy consultations for participants in this group will last 30 minutes initially and then 20 minutes thereafter, consistent with clinical practice. Physiotherapists will prescribe 5-6 strengthening exercises from a pre-determined list to be performed at home three times/week, including two quadriceps exercises, one each for hip abductors, hamstrings and calf, and any other as appropriate and a personalised physical activity plan.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Diet plus exercise — The diet program has two phases: 1) intensive weight loss through a ketogenic very low calorie diet VLCD, and 2) transition from ketogenic VLCD onto a healthy eating plan for weight maintenance. Meal replacements will be provided to participants free of charge from the start of the trial to a maximum of 14 weeks (12 weeks for the ketogenic diet and 2 weeks for transition). If a participant does not wish to transition off the ketogenic diet after 14 weeks but wants to continue or if they wish to recommence the ketogenic diet any time after week 14 they will need to purchase meal replacements themselves at their own cost.
  Participants will be encouraged to aim to lose at least 10% body weight.
  Arms: Diet plus exercise
Other: Exercise — The trial coordinator will have provided participants with educational material about OA, handouts of home exercises including photographs and descriptions, a logbook for recording home program completion and resistance exercise bands ahead of their first appointment. Physiotherapists will prescribe 5-6 strengthening exercises from a pre-determined list to be performed at home three times/week, including two quadriceps exercises, one each for hip abductors, hamstrings and calf, and any other as appropriate. Review and modification will occur at each consultation to maintain moderate intensity (effort of ≥5 out of 10 (hard) on a modified Borg Rating of Perceived Exertion scale). The physiotherapist will also prescribe a personalised physical activity plan in collaboration with the participant that is supported and progressed over time.

SUMMARY:
The aim of this randomized controlled trial is to evaluate the effects of a physiotherapist-delivered dietary weight loss program on clinical outcomes among people with knee osteoarthritis (OA) who have overweight or obesity. The primary hypothesis is that a physiotherapist-delivered dietary weight loss plus exercise program will be more effective in achieving weight loss than a physiotherapist-delivered exercise program alone. Approximately 6-9 physiotherapists in Melbourne, Australia will be recruited and trained in weight management for OA patients, as well as trained in how to deliver the specific study interventions. The same therapists will deliver the intervention in both arms of the trial. 88 participants with knee OA will be recruited from the community and randomized into one of the two arms a) diet plus exercise intervention or b) exercise intervention alone. Participants in both groups will be asked to attend 6 consultations with the physiotherapist over 6 months. Questionnaire and laboratory-based outcome measures will be completed by participants at baseline and at the end of the 6 month intervention period. A biostatistician will analyse blinded, de-identified data.

DETAILED DESCRIPTION:
Clinical guidelines for the management of knee OA recommend exercise as a core treatment for all patients as well as losing weight for those patients who also have overweight/obesity. However, health care systems are frequently under strain often experiencing limited numbers of, and access to, clinicians with specialist weight loss and health behavior change skills. New models of care for OA are needed that support expanded practice roles for clinicians. Physiotherapists are key providers of exercise therapy for knee OA but the effectiveness of physiotherapists to deliver a dietary weight loss program for patients with knee OA is not known.

This study is a randomized controlled trial for which the aim is to evaluate the effects of a physiotherapist-delivered dietary weight loss program in addition to exercise, on weight loss and other clinical outcomes among people with knee OA who have overweight or obesity. The research question is: Is a 6-month physiotherapist-delivered dietary weight loss plus exercise program more effective for improving clinical outcomes than a physiotherapist-delivered exercise program alone in people with knee OA who have overweight or obesity?

Clinical practice guidelines for knee OA recommend patients who have overweight or obesity should lose at least 5-7.5% of body weight. Therefore the study is powered to detect a conservative between-group difference in weight loss of 5% of body weight assuming no change in weight in the control group (exercise only) based on previous research.

A total of 88 participants with chronic knee pain and a clinical diagnosis of knee OA will be recruited from the community. Participants will be enrolled into the study following informed consent and completion of baseline questionnaires and laboratory-based measures. Each participant will be randomly allocated to receive a: a) diet plus exercise program or; b) exercise program alone, over 6 months.

The randomization schedule will be computer generated and prepared by the biostatistician (permuted block sizes 6 to 12) stratified by physiotherapist and sex of participant. The schedule will be stored on a password-protected website maintained by a researcher not involved in either participant recruitment or administration of outcome measures. Group allocation will be revealed to the physiotherapists and the participants by this same researcher following randomisation.

The physiotherapists will undertake comprehensive training prior to being allocated trial participants. Physiotherapists will be trained in weight management, the ketogenic very low calorie diet and trial procedures.

Study participants in both groups will visit a physiotherapist in-person for six individual sessions over 6 months. Participants will choose the therapist according to location. The same therapist will undertake all consultations with any given participant.

Those in the diet plus exercise group will undertake a ketogenic very low calorie diet (VLCD) which has been demonstrated as a safe and effective means of achieving rapid weight loss in the adult population with overweight/obesity. They will receive meal replacements (maximum 2 per day) for up to 14 weeks from the start of the study as well as educational resources. Both groups will also undertake a home-based lower limb muscle strengthening exercise and physical activity program.

A biostatistician will analyse blinded data. Comparative analyses between groups will use intention-to-treat. Multiple imputation will be used to account for missing data if the proportion of missing data is >5%. For the primary outcome, the difference in mean percentage change in body weight will be compared between groups using mixed linear regression model adjusting for baseline weight and the stratification variables, with random intercepts for treating physiotherapist. Similar analyses will be conducted for continuous secondary outcomes. We will also calculate the proportion of participants achieving ≥5% and ≥10% loss of body weight in both groups. For binary outcomes, logistic regression models will be fit using generalized estimating equations, with risk differences and 95% confidence intervals calculated.

ELIGIBILITY:
Inclusion Criteria:

* Meet the National Institute for Health and Care Excellence [47] clinical criteria for OA: age≥45 years; activity-related knee joint pain; morning knee stiffness ≤ 30 mins
* report history of knee pain ≥ 3 months
* report knee pain on most days of the past month
* report a minimum knee pain score of 4 on an 11-point numeric rating scale during walking over the previous week
* body mass index (BMI) >27 kg/m2
* those using hypertensive medication must be willing to have their blood pressure checked (this can be self-monitoring, at a pharmacist or at a GP) if they feel light-headed or dizzy at any point during the study
* able to give informed consent and to participate fully in the interventions and assessment procedures

Exclusion Criteria:

* weight >150 kgs (due to the added complexities of additional nutritional requirements for individuals above this weight)
* inability to speak English
* on waiting list for/planning knee/hip surgery or bariatric surgery in next 6 months
* arthroplasty on affected knee
* recent knee surgery on affected knee (past 6 months);
* self-reported inflammatory arthritis (e.g. rheumatoid arthritis)
* weight loss of > 2 kg over the previous 3 months
* already actively trying to lose weight by any of the following mechanisms:using meal replacements for weight loss; being a member of a slimming club (e.g. weight watchers); receiving support from another health care professional for weight loss; using any drugs prescribed to aid in weight loss; using structured meal programs for weight loss such as 'Lite n' Easy'
* unwilling to continue current dietary patterns if randomized to exercise only group
* unable to undertake ketogenic VLCD for medical reasons including self-reported: diagnosis of Type 1 diabetes;Type 2 diabetes requiring insulin or other medication apart from metformin; Warfarin use; stroke or cardiac event in previous 6 months; unstable cardiovascular conditions; fluid intake restrictions; renal (kidney) problems (unless clearance is obtained from a general practitioner (GP), including GP confirmation that estimated glomerular filtration rate >30 mL/min/1.73m2); any neurological condition affecting lower limbs; vegan dietary requirements due to complexity of delivering a nutritionally complete diet within the ketogenic diet regime

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Body weight | Change between baseline and 6 months post randomization
  Measured using calibrated digital laboratory platform scales (TCS-2 series) to 2 decimal places, the percentage of body weight change (baseline-follow up/baseline x100%) will be calculated as the primary outcome

SECONDARY OUTCOMES:
Body mass index (BMI) | Change between baseline and 6 months post randomization
  Calculated from height and weight, in Kg/m2
Waist circumference | Change between baseline and 6 months post randomization
  Measured according to standardised instructions using a tape measure in centimetres to 1 decimal place
Waist to hip ratio | Change between baseline and 6 months post randomization
  Measured according to standardized instructions using a tape measure and presented as a ratio
Severity of knee pain during walking | Change between baseline and 6 months post randomization
  Scored on an 11-point NRS for average knee pain during walking in the last week, Ranges from 0 to 10; where 0=no pain and 10=worst pain possible
Intermittent and constant osteoarthritis pain measure (iCOAP) | Change between baseline and 6 months post randomization
  11-item tool with constant and intermittent pain subscales. Ranges from 0 to 20 for constant pain subscale and 0 to 24 for intermittent subscale and 0 to 44 for total score with 44 being maximal pain
Physical function subscale of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Change between baseline and 6 months post randomization
  Scored using 17 questions regarding knee function in the last 48 hours, with Likert response options ranging from no dysfunction to extreme dysfunction. Ranges from 0 (no dysfunction) to 68 (maximum dysfunction)
Global overall improvement in knee problems | 6 months post randomization
  Scored using a 7-point global rating of change Likert scale from with response options ranging from "much worse" to "much better" when compared to baseline. Participants who indicate that they are "moderately better" or "much better" will be classified as improved. All other respondents will be classified as not improved
Quality of life (AQoL-6D) | Change between baseline and 6 months post randomization
  Scored using the 20-item Assessment of Quality of Life II Instrument (6D version), which covers the topics of Independent Living, Relationships, Mental Health, Coping, Pain and Senses to come up with one overall value representing quality of life. Total score ranges from -0.04 to 1.00; higher scores indicate better quality of life
Physical Activity scale for the elderly (PASE) | Change between baseline and 6 months post randomization
  Scored via 10 questions about frequency and duration of recreational, household and occupational physical activity undertaken over the past 7 days. Scores range from 0 to 400+; higher scores indicate greater levels of physical activity
30 sec chair stand test | Change between baseline and 6 months post randomization
  Number of complete chair stands completed in 30 secs. Greater number indicates better function
40 m fast paced walk test | Change between baseline and 6 months post randomization
  Time to taken to walk 4 x 10 m quickly but safely. Measured in Metres/Second. Greater speed indicates better function
Stair climb test | Change between baseline and 6 months post randomization
  Time taken for participant to ascend and descend a flight of stairs. Measured in seconds, shorter time indicates better function
Quadriceps muscle strength | Change between baseline and 6 months post randomization
  Maximum voluntary isometric strength will be assessed using an isokinetic dynamometer with the knee at 60 degrees knee flexion. Peak torque over 3 maximal efforts lasting 3 seconds will be recorded. Measured in Nm/kg
Weight Self-Stigma Questionnaire (WSSQ) | Change between baseline and 6 months post randomization
  Self-reported and scored on a 12-item questionnaire, with two 6-item sub-scales. Each item rated on a 5-point Likert scale where from 1=completely disagree to 5=completely agree. Total and subscale scores will be reported with higher scores indicating greater internalized weight stigma.
Self-efficacy for eating control | Change between baseline and 6 months post randomization
  Weight Efficacy Lifestyle (WEL) Questionnaire Short Form. Scored from 8 statements regarding eating control on a 10-point NRS where 0="Not confident at all that I can resist the desire to eat" and 9="Very confident that I can resist the desire to eat". The WEL Short Form is validated to the original 20 item WEL which was based on 5 constructs [44]: negative emotions, availability, social pressure, physical discomfort, and positive activities. Total scores range from 0-80; higher scores indicate greater eating self-efficacy
Arthritis self-efficacy scale | Change between baseline and 6 months post randomization
  Arthritis self-efficacy scale short form. Scored from 8 questions on a 10-point NRS where 1="Very uncertain" and 10="Very certain". The scale assess self-efficacy for control of pain, physical function and frustration associated with OA. Scores are the mean of the items in each scale. Total scores are an average of the 8 items with a range from 1 to 10; higher scores indicate higher self-efficacy.

OTHER OUTCOMES:
Adverse events | 6 months post randomization
  Self-reported - Number of participants who experience adverse events, number of adverse events, type of adverse events and actions taken in response to adverse events, relatedness to the intervention
Attendance at consultations | Throughout intervention period (0-6 months)
  Recorded by physiotherapist for each consultation, number of consultations attended recorded
Duration of consultations | Throughout intervention period (0-6 months)
  Taken from physiotherapist treatment records
Physiotherapist contact with study investigators for advice or support relating to the weight loss program during delivery of the intervention | Throughout intervention period (0-6 months)
  Taken from study investigator records, the number of physiotherapists who contacted study investigators, number of contacts and the reasons for contact will be recorded
Adherence with strengthening exercise program | 6 months post randomization
  Self-reported number of exercise sessions in the last 2 weeks (options of 0, 1,2,3,4,5 and 6). Taken from a range from 0-6 sessions, converted to a % out of the 6 prescribed sessions.
Rating of adherence with strengthening exercise program Rating of adherence with strengthening exercise program Rating of adherence with strengthening exercise program | 6 months post randomization
  Self-reported and scored on a 11-point NRS for "I have been doing my exercise sessions the number of times I was asked to by my POWER physiotherapist (e.g. three times per week)" over the previous 6 months. Ranges from 0 to 10; where 0=strongly disagree and 10=strongly agree
Adherence with physical activity plan | 6 months post randomization
  Self-reported and scored on a 11-point NRS for "I followed the physical activity plan that my POWER trial physiotherapist helped me to develop" over the previous 6 months. Ranges from 0 to 10; 0=strongly disagree and 10=strongly agree
Adherence with diet program (diet plus exercise group only) | 6 months post randomization
  Self-reported and scored on a 11-point NRS for "I followed the diet plan as it was outlined by my POWER trial physiotherapist" over the previous 6 months. Ranges from 0 to 10; 0=strongly disagree and 10=strongly agree
Number of weeks participants used meal replacements (diet plus exercise group only) | 6 months post randomization
  Self-reported, number (0-24)
Satisfaction with the allocated program | 6 months post randomization
  Scored on a 7-point global rating of change scale with response options from "extremely dissatisfied" to "extremely satisfied". Participants indicating, they are "moderately satisfied" or "extremely satisfied" will be classified as satisfied with the program
Working Alliance Inventory Short Revised | 6 months post randomization for patients, and at consultation 4 and 6 for physiotherapists
  Self-reported by both patients and physiotherapists. 12-item questionnaire which measures the strength of the therapeutic alliance A 7-point Likert Scale is used for each question. Overall scores range from 12 to 84 (with higher scores indicating a stronger therapeutic alliance).
Co-intervention use | Baseline and 6 months post randomization
  Self-reported. Participants will complete a table listing different co-interventions used to manage their knee condition and their weight in the previous 3 months. Number of co-interventions and number of participants using co-interventions.
Medication use | Baseline and 6 months post randomization
  Self-reported. Participants will complete a table detailing a variety of pain and arthritis medications and supplements used in the previous month.
Attitudes towards different health care practitioners' delivery of weight loss intervention | Change between baseline and 6 months post randomization
  Self-reported. Participants will rate their confidence in 3 different health care practitioners delivering weight loss interventions by responding to the statement 'I am confident that a [general practitioner / dietician / physiotherapist] could deliver a dietary weight loss program' A 5-point Likert Scale is used for each health practitioner, 1=strongly disagree, to 5=strongly agree. Each practitioner will receive a score from 1-5 with higher scores indicating higher confidence in the practitioner's ability to deliver weight loss intervention
Attitudes and experiences of participants to the physiotherapist delivered diet program (diet plus exercise group only) | 6 months post randomization
  Self-reported. Participants will respond to a series of 8 custom statements exploring their perception of the knowledge and skills of their physiotherapist and their confidence in, and comfort working with, the physiotherapist for delivery and support of a dietary weight loss program. A 5-point Likert Scale is used for each question, anchored at '1'=strongly disagree, to '5'=strongly agree. Scores range from 1-5 for each statement

CONTACTS AND LOCATIONS:
Overall Officials: Kim Bennell, PhD, Principal Investigator — University of Melbourne
Locations (1):
- University of Melbourne, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: We will share all data that support results of the trial following publication. Additional data that have not been published will be withheld until at least six months after publication.
Access Criteria: Data will be made available as required for specific, approved analyses. Data will be provided from locked, cleaned, and de- identified study database. All requests for data sharing will be reviewed by the Principal Investigator to ensure no conflict with any planned sub analyses and to ensure that the data are shared in an ethical and protected manner. Analyses for non-commercial purposes are eligible. Before any analysis, a signed Confidentiality Agreement and/or Data Sharing Agreement is required.

REFERENCES:
- [Derived] Allison K, Jones S, Hinman RS, Pardo J, Li P, DeSilva A, Quicke JG, Sumithran P, Prendergast J, George E, Holden MA, Foster NE, Bennell KL. Alternative models to support weight loss in chronic musculoskeletal conditions: effectiveness of a physiotherapist-delivered intensive diet programme for knee osteoarthritis, the POWER randomised controlled trial. Br J Sports Med. 2024 May 2;58(10):538-547. doi: 10.1136/bjsports-2023-107793. PMID 38637135
- [Derived] Bennell KL, Jones SE, Hinman RS, McManus F, Lamb KE, Quicke JG, Sumithran P, Prendergast J, George ES, Holden MA, Foster NE, Allison K. Effectiveness of a telehealth physiotherapist-delivered intensive dietary weight loss program combined with exercise in people with knee osteoarthritis and overweight or obesity: study protocol for the POWER randomized controlled trial. BMC Musculoskelet Disord. 2022 Jul 30;23(1):733. doi: 10.1186/s12891-022-05685-z. PMID 35907828